CLINICAL TRIAL: NCT05145699
Title: A Pilot Study on the Feasibility Study of a Novel VR-based Post-stroke Hemineglect Evaluation System
Brief Title: A Pilot Study on the Feasibility Study of a Novel Virtual Reality (VR)-Based Post-stroke Hemineglect Evaluation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: B-2108-705-302
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Complication
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Right hemispheric stroke with hemineglect (Experimental)
  Interventions: Device: VR-based post-stroke hemineglect evaluation system
- Right hemispheric stroke without hemineglect (Active Comparator)
  Interventions: Device: VR-based post-stroke hemineglect evaluation system
- Normal people (Other)
  Interventions: Device: VR-based post-stroke hemineglect evaluation system

INTERVENTIONS:
Device: VR-based post-stroke hemineglect evaluation system — Evaluation system applied with virtual environment using Pico Neo 2 eye

SUMMARY:
The normal value of the new virtual reality (VR)-based hemineglect evaluation system is obtained and its validity is checked by whether there is a difference in the evaluation results between normal people, stroke patients with hemineglect, and stroke patients without hemineglect. And, the usability of the virtual reality-based hemineglect evaluation system is confirmed.

DETAILED DESCRIPTION:
This pilot study included 50 stroke patients with right hemisphere lesion and 25 healthy people.

The normal value for each item is determined based on the result value for each item of the virtual reality (VR)-based hemineglect evaluation system in normal people.

It is checked whether there is a difference in the results measured using the VR-based hemineglect evaluation system in normal persons, stroke patients with hemineglect, and stroke patients without hemineglect.

Structural validity is confirmed by examining the correlation between the measured values of the virtual VR-based hemineglect evaluation system and Korean Version of Modified Barthel Index (K-MBI), Mini Mental State Examination (MMSE), and Behavioral Inattention Test-Conventional (BIT-C) in stroke patients with hemineglect.

Check the required time and test stability of the evaluation using the VR-based hemineglect evaluation system.

ELIGIBILITY:
Inclusion Criteria:

(Stroke patients)

* Right handed
* Patients with first onset stroke, with right brain lesions confirmed by imaging tests (MRI, CT)
* Onset of stroke more than 1week (Normal people)
* Right handed
* Who has no problem in identifying objects with wearing VR head gear.

Exclusion Criteria:

(Stroke patients)

* Patients with unilateral neglect due to other causes.
* Patients with neurological diseases other than stroke (Parkinson's disease, Alzheimer's disease, etc.)
* Patients with severe cognitive impairment.
* Patients with underlying diseases or medical history that may cause visual impairment.

(Normal people)

* Who has a neurological disease such as stroke, traumatic brain injury, Parkinson's disease, or Alzheimer's disease.
* Who has a severe cognitive impairment.
* Who has a underlying diseases or medical history that may cause visual impairment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
8 items of virtual reality-based hemineglect evaluation system | up to 1 year
  (1)Visual extinction, (2)Visual tracking, (3-6)Visual scanning, (7)Auditory, (8)Activities of Daily Living (ADL)

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, Ph.D, Principal Investigator — Seoul National University Bundang Hospital, Seongnam, South Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided